CLINICAL TRIAL: NCT06007404
Title: The Role of Circulating Meta-Inflammatory Monocytes in Adolescent Insulin Resistance
Brief Title: Understanding Metabolism and Inflammation Risks for Diabetes in Adolescents
Status: Recruiting | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kanakadurga Singer, Associate Professor, University of Michigan
Other Study IDs: HUM00208301; R01DK130864 (NIH)
Record Dates: First submitted 2023-06-10; First posted 2023-08-23 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes; Insulin Resistance; Obesity; Metabolic Disease; PreDiabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Obesity; Metabolic Diseases; Prediabetic State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Normal weight: BMI ≥ 5th percentile & < 85th percentile
- Obese weight: BMI ≥ 95th percentile
- PreDiabetes: HbA1c > 5.7%
- Type 2 Diabetes: Diagnosed with Type 2 Diabetes
- Overweight: BMI > 86th percentile and <94th percentile

SUMMARY:
This research study collects health-related information and blood samples to better understand how body composition, lifestyle habits, and diet influence meta-inflammatory monocytes (MiMos) in adolescents. The hypothesis of this study is that adolescents at risk for metabolic disease have enhanced MiMo related activities leading to insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Between 14 and 18 years of age
* Tanner stage 4 or 5 (mature adult stage of puberty)
* Normal weight (BMI ≥ 5th percentile & < 85th percentile), overweight (BMI > 86th percentile) & < 94th percentile), obese weight (BMI percentile ≥ 95th percentile), and/or pre-diabetes (HbA1c > 5.7%)
* For Type 2 Diabetes cohort, diagnosis of Type 2 Diabetes

Exclusion Criteria:

* Currently pregnant
* Use medications known to affect glucose metabolism (immunosuppressive medications, cancer medications, or high dose steroids), unless prescribed for Type 2 Diabetes management
* Prior diagnosis of autoimmune disease, cancer, or a cognitive or perceptual disability that would inhibit following directions of study staff
* Allergies or intolerance to milk, soy, or palm oil

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants may be recruited from a variety of sites including University of Michigan clinical sites, non-University of Michigan clinical sites, local communities and schools throughout Southeast Michigan, and the University of Michigan campus.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Glucose (OGTT) | 120 minutes
  Plasma Glucose (mg/dL) will be measured prior to, and throughout, an Oral Glucose Tolerance Test (OGTT). Measurements will be taken at baseline (fasting) and 30, 60, 90 and 120 minutes after consumption of glucose dose
Insulin (OGTT) | 120 minutes
  Plasma Insulin (µU/mL) will be measured prior to, and throughout, an Oral Glucose Tolerance Test (OGTT). Measurements will be taken at baseline (fasting) and 30, 60, 90 and 120 minutes after consumption of glucose dose
Glucose (MMTT) | 180 minutes
  Plasma Glucose (mg/dL) will be measured prior to, and throughout, a Mixed Meal Tolerance Test (MMTT). Measurements will be taken at baseline (fasting) and 30, 60, 90, 120 and 180 minutes after consumption of high fat shake.
Insulin (MMTT) | 180 minutes
  Plasma Insulin (µU/mL) will be measured prior to, and throughout, a Mixed Meal Tolerance Test (MMTT). Measurements will be taken at baseline (fasting) and 30, 60, 90, 120 and 180 minutes after consumption of high fat shake.
Monocyte /macrophage populations by flow cytometry | 180 minutes
  Frequencies by flow cytometry. Measurements will be taken at baseline sample and 180 minutes after consumption of high fat shake

SECONDARY OUTCOMES:
Free fatty acids (MMTT) | 180 minutes
  Serum Free fatty acids (mmol/L) will be measured prior to, and throughout, a Mixed Meal Tolerance Test (MMTT). Measurements will be taken at baseline (fasting) and 30, 60, 90, 120 and 180 minutes after consumption of high fat shake
Triglycerides (MMTT) | 180 minutes
  Serum Triglycerides (mg/dL) will be measured prior to, and throughout, a Mixed Meal Tolerance Test (MMTT). Measurements will be taken at baseline (fasting) and 30, 60, 90, 120 and 180 minutes after consumption of high fat shake

CONTACTS AND LOCATIONS:
Overall Officials: Kanakadurga Singer, MA, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Genomic and associated phenotypic data will be shared through NIH-designated data repositories.
Supporting Information: Study Protocol
Time Frame: Genotype/sequencing and phenotype data will be submitted after the genotyping/sequencing data have been cleaned. Following submission, data will be released within six months.
Access Criteria: In regards to genomic data, individual-level data will be deidentified and made available through controlled-access.